CLINICAL TRIAL: NCT06560008
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of EnXtra® and EnXtra® + Caffeine on Mental Alertness and Fatigue in Healthy Individuals
Brief Title: A Study to Evaluate the Effect of EnXtra® and EnXtra® + Caffeine on Mental Alertness and Fatigue in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Enovate Biolife Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: EB/240403/ENXTRA/CSF
Record Dates: First submitted 2024-08-08; First posted 2024-08-19 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Fatigue; Mental Alertness
MeSH Terms: conditions — Fatigue | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Acute stage: Randomized, double-blind, placebo-controlled, single-dose, 4-way, cross-over, study Sub-Acute Stage: Randomized, double-blind, placebo-controlled, 4 arms, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EnXtra® (300 mg) + Placebo (300 mg) (Active Comparator): Acute Stage: Two capsules to be taken after breakfast orally 1 (single dose) x 4 periods = 4 days Sub-acute Stage: Two capsules to be taken after breakfast orally once a day for 28 days
  Interventions: Dietary Supplement: EnXtra® (300 mg) + Placebo (300 mg)
- Caffeine (200 mg) + Placebo (300 mg) (Active Comparator): Acute Stage: Two capsules to be taken after breakfast orally 1 (single dose) x 4 periods = 4 days Sub-acute Stage: Two capsules to be taken after breakfast orally once a day for 28 days
  Interventions: Dietary Supplement: Caffeine (200 mg) + Placebo (300 mg)
- EnXtra® (300 mg) + Caffeine (200 mg) (Active Comparator): Acute Stage: Two capsules to be taken after breakfast orally 1 (single dose) x 4 periods = 4 days Sub-acute Stage: Two capsules to be taken after breakfast orally once a day for 28 days
  Interventions: Dietary Supplement: EnXtra® (300 mg) + Caffeine (200 mg)
- Placebo (MCC 300 mg) + Placebo (300 mg) (Placebo Comparator): Acute Stage: Two capsules to be taken after breakfast orally 1 (single dose) x 4 periods = 4 days Sub-acute Stage: Two capsules to be taken after breakfast orally once a day for 28 days
  Interventions: Dietary Supplement: Placebo (MCC 300 mg) + Placebo (300 mg)

INTERVENTIONS:
Dietary Supplement: EnXtra® (300 mg) + Placebo (300 mg) — Two capsules to be taken after breakfast orally once a day (4 single doses in Acute stage and for 28 days in sub-acute stage)
  Arms: EnXtra® (300 mg) + Placebo (300 mg)
Dietary Supplement: Caffeine (200 mg) + Placebo (300 mg) — Two capsules to be taken after breakfast orally once a day (4 single doses in Acute stage and for 28 days in sub-acute stage)
  Arms: Caffeine (200 mg) + Placebo (300 mg)
Dietary Supplement: EnXtra® (300 mg) + Caffeine (200 mg) — Two capsules to be taken after breakfast orally once a day (4 single doses in Acute stage and for 28 days in sub-acute stage)
  Arms: EnXtra® (300 mg) + Caffeine (200 mg)
Dietary Supplement: Placebo (MCC 300 mg) + Placebo (300 mg) — Two capsules to be taken after breakfast orally once a day (4 single doses in Acute stage and for 28 days in sub-acute stage)
  Arms: Placebo (MCC 300 mg) + Placebo (300 mg)

SUMMARY:
Acute Stage: The present study is a randomized, double-blind, placebo-controlled, single-dose, 4-way, cross-over, study. Approximately not more than 170 individuals will be screened and considering a screening failure rate of 25%, approximately 128 individuals will be randomized in a ratio of 1:1:1:1 to receive one of the IPs and will be assigned a unique randomization code. In this stage, approximately 114 individuals will complete the study, after accounting for a dropout/withdrawal rate of 15%. The intervention duration is 4 days [1 (single dose) x 4 periods].

Sub-Acute Stage: The present study is a randomized, double-blind, placebo-controlled, 4 arms, parallel study. In this stage, approximately 112 individuals will be re-randomized in a ratio of 1:1:1:1 to receive one of the IPs and will be assigned a unique randomization code. Each group will have not less than 24 completed participants after accounting for a dropout/withdrawal rate of 15%. The intervention duration is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 40 years.
* Individuals who have night sleep of 8±1 hours.
* Individuals with BMI ≥ 18 and ≤ 29.9 kg/meter square
* Alertness score (Jin Fan's ANT) of 50±20 ms after 24 hours of caffeine abstinence.
* Individuals habituated to have at least 2 cups of coffee in a day.
* Individuals with a feeling of sleepiness having Karolinska Sleepiness Scale (KSS) of more than 7 during caffeine abstinence.
* Individuals who fit in physical examination, vital signs and all screening tests are within acceptable limits, according to the physician/investigator's opinion.
* Individuals having computer literacy to perform the required assessments.
* Individuals willing to provide signed consent.

Exclusion Criteria:

* Individuals diagnosed with sleep disorders secondary to another health problem.
* Individuals with a trait of excessive food cravings.
* History of consumption of psychedelic drugs.
* Individuals who are caffeine dependent i.e. having a history of more than 3 cups (≥200 ml) in a day.
* Individuals taking energy/ cognitive/ sedative supplements and are unwilling to stop taking those supplements for the duration of the study period.
* Recent history of physical, emotional, and social trauma within the last three months.
* Individuals who consume pain-relieving medications more than once per week.
* Use of the following medications during the study period: oral or injectable corticosteroid, sedating antihistamines (e.g. cold, allergy, motion sickness), psychotropic medications or hypnotics, benzodiazepine, narcotics, or any illicit drugs.
* Gastrointestinal, hepatic, respiratory, psychiatric, kidney, or cardiovascular disorder (<3 months before inclusion).
* Recent (<3 months before inclusion) change in lifestyle (food, body weight, sport, drug, and dietary supplement).
* Addiction or history of substance abuse.
* Consumption of more than 3 units of alcohol per day. (one unit is equal to 45 ml of hard liquor, 150 ml of wine or a pint of beer)
* Abnormal Thyroid Stimulating Hormone (TSH) value which is less than 0.40 or more than 5.0 μIU/mL.
* Known Diabetics.
* Hypertensives defined as SBP more than 140 mm Hg and/or DBP more than 90 mm Hg with or without anti-hypertensives.
* Use another investigational product within 90 days of the screening visit.
* Individuals with a history of or complications from malignant tumors.
* History of any significant neurological and psychiatric condition that may affect the participation and inference of the study's endpoints.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Any condition that could, in the opinion of the investigator, preclude the individual's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
To determine the effect of EnXtra® and EnXtra® + Caffeine on alertness score as assessed by the change in the Jin Fan Alertness score as compared to placebo and caffeine in Acute stage. | Day 0 at 0, 1, 3 and 5 hours ± 15 minutes post IP
  The Attention Network Test (ANT) is an assessment tool to evaluate efficacy of three distinct attention networks: alerting, orienting, and executive networks.
  Alerting effect = mean Response Time (RT) (correct no cue) - mean RT (correct centre cue) Orienting effect = mean RT (correct centre cue) - mean RT (correct spatial cue) Conflict effect = mean RT (correct incongruent) - mean RT (correct congruent) Correct: correctness of response No cue condition: participant does not receive any cue before the target stimulus appears.
  Spatial cue is usually presented in the form of an arrow, pointing in the location where the target stimulus will show up.
  Centre cue condition, A cue appears at the screen's center just before the target stimulus.
  Incongruent: The target stimulus is flanked by distractors oriented in the opposite direction.
  Congruent: The target stimulus is flanked by distractor stimuli oriented in the same direction.
To determine the effect of EnXtra® and EnXtra® + Caffeine on alertness score as assessed by the change in the Jin Fan Alertness score as compared to placebo and caffeine in Acute stage. | Day 5 at 0, 1, 3 and 5 hours ± 15 minutes post IP
  The Attention Network Test (ANT) is an assessment tool to evaluate efficacy of three distinct attention networks: alerting, orienting, and executive networks.
  Alerting effect = mean Response Time (RT) (correct no cue) - mean RT (correct centre cue) Orienting effect = mean RT (correct centre cue) - mean RT (correct spatial cue) Conflict effect = mean RT (correct incongruent) - mean RT (correct congruent) Correct: correctness of response No cue condition: participant does not receive any cue before the target stimulus appears.
  Spatial cue is usually presented in the form of an arrow, pointing in the location where the target stimulus will show up.
  Centre cue condition, A cue appears at the screen's center just before the target stimulus.
  Incongruent: The target stimulus is flanked by distractors oriented in the opposite direction.
  Congruent: The target stimulus is flanked by distractor stimuli oriented in the same direction.
To determine the effect of EnXtra® and EnXtra® + Caffeine on alertness score as assessed by the change in the Jin Fan Alertness score as compared to placebo and caffeine in Acute stage. | Day 10 at 0, 1, 3 and 5 hours ± 15 minutes post IP
  The Attention Network Test (ANT) is an assessment tool to evaluate efficacy of three distinct attention networks: alerting, orienting, and executive networks.
  Alerting effect = mean Response Time (RT) (correct no cue) - mean RT (correct centre cue) Orienting effect = mean RT (correct centre cue) - mean RT (correct spatial cue) Conflict effect = mean RT (correct incongruent) - mean RT (correct congruent) Correct: correctness of response No cue condition: participant does not receive any cue before the target stimulus appears.
  Spatial cue is usually presented in the form of an arrow, pointing in the location where the target stimulus will show up.
  Centre cue condition, A cue appears at the screen's center just before the target stimulus.
  Incongruent: The target stimulus is flanked by distractors oriented in the opposite direction.
  Congruent: The target stimulus is flanked by distractor stimuli oriented in the same direction.
To determine the effect of EnXtra® and EnXtra® + Caffeine on alertness score as assessed by the change in the Jin Fan Alertness score as compared to placebo and caffeine in Acute stage. | Day 15 at 0, 1, 3 and 5 hours ± 15 minutes post IP
  The Attention Network Test (ANT) is an assessment tool to evaluate efficacy of three distinct attention networks: alerting, orienting, and executive networks.
  Alerting effect = mean Response Time (RT) (correct no cue) - mean RT (correct centre cue) Orienting effect = mean RT (correct centre cue) - mean RT (correct spatial cue) Conflict effect = mean RT (correct incongruent) - mean RT (correct congruent) Correct: correctness of response No cue condition: participant does not receive any cue before the target stimulus appears.
  Spatial cue is usually presented in the form of an arrow, pointing in the location where the target stimulus will show up.
  Centre cue condition, A cue appears at the screen's center just before the target stimulus.
  Incongruent: The target stimulus is flanked by distractors oriented in the opposite direction.
  Congruent: The target stimulus is flanked by distractor stimuli oriented in the same direction.
To determine the effect of EnXtra® and EnXtra® + Caffeine on alertness score as assessed by the change in the Jin Fan Alertness score as compared to placebo and caffeine in Sub-acute stage. | Day 20 at 0 hours post IP
  The Attention Network Test (ANT) is an assessment tool to evaluate efficacy of three distinct attention networks: alerting, orienting, and executive networks.
  Alerting effect = mean Response Time (RT) (correct no cue) - mean RT (correct centre cue) Orienting effect = mean RT (correct centre cue) - mean RT (correct spatial cue) Conflict effect = mean RT (correct incongruent) - mean RT (correct congruent) Correct: correctness of response No cue condition: participant does not receive any cue before the target stimulus appears.
  Spatial cue is usually presented in the form of an arrow, pointing in the location where the target stimulus will show up.
  Centre cue condition, A cue appears at the screen's center just before the target stimulus.
  Incongruent: The target stimulus is flanked by distractors oriented in the opposite direction.
  Congruent: The target stimulus is flanked by distractor stimuli oriented in the same direction.
To determine the effect of EnXtra® and EnXtra® + Caffeine on alertness score as assessed by the change in the Jin Fan Alertness score as compared to placebo and caffeine in Sub-acute stage. | Day 48 at 1, 3 and 5 hours ± 15 minutes post IP
  The Attention Network Test (ANT) is an assessment tool to evaluate efficacy of three distinct attention networks: alerting, orienting, and executive networks.
  Alerting effect = mean Response Time (RT) (correct no cue) - mean RT (correct centre cue) Orienting effect = mean RT (correct centre cue) - mean RT (correct spatial cue) Conflict effect = mean RT (correct incongruent) - mean RT (correct congruent) Correct: correctness of response No cue condition: participant does not receive any cue before the target stimulus appears.
  Spatial cue is usually presented in the form of an arrow, pointing in the location where the target stimulus will show up.
  Centre cue condition, A cue appears at the screen's center just before the target stimulus.
  Incongruent: The target stimulus is flanked by distractors oriented in the opposite direction.
  Congruent: The target stimulus is flanked by distractor stimuli oriented in the same direction.

SECONDARY OUTCOMES:
To determine the effect of EnXtra® and EnXtra® + Caffeine on Eye-hand coordination as assessed by Nine hole peg test (NHPT) as compared to placebo and caffeine in Acute stage. | Day 0; Day 5; Day 10; Day 15 - 0, 1, 3 & 5 hours ±15 minutes post IP
  The NHPT assesses eye-hand coordination in individuals. This study focuses on the dominant hand's performance.
  Metrics recorded for assessment:
  Moving Duration - 1: Time to move the first peg from the holder to the board, indicating initial movement speed and fluidity.
  First Peg Selection - 1: Time from the start of the test until the first peg is picked up, indicating readiness and initial response speed.
  Transport Drops - 1: Number of times the first peg is dropped during transport, assessing precision and control.
  Moving Duration - 2: Similar to Moving Duration - 1 for the second peg, providing insight into consistency and endurance over multiple attempts.
  First Peg Selection - 2: Time taken to select the first peg again, measuring sustained attention and readiness.
  Transport Drops - 2: No. of drops during the second transport attempt, evaluating precision and control.
  An increase in moving duration indicates a decline in eye-hand coordination speed.
To determine the effect of EnXtra® and EnXtra® + Caffeine on Eye-hand coordination as assessed by Nine hole peg test (NHPT) as compared to placebo and caffeine in Sub-acute stage. | Day 20 - 0 hours, Day 48 - 1, 3 & 5 hours ±15 minutes post IP
  The NHPT assesses eye-hand coordination in individuals. This study focuses on the dominant hand's performance.
  Metrics recorded for assessment:
  Moving Duration - 1: Time to move the first peg from the holder to the board, indicating initial movement speed and fluidity.
  First Peg Selection - 1: Time from the start of the test until the first peg is picked up, indicating readiness and initial response speed.
  Transport Drops - 1: Number of times the first peg is dropped during transport, assessing precision and control.
  Moving Duration - 2: Similar to Moving Duration - 1 for the second peg, providing insight into consistency and endurance over multiple attempts.
  First Peg Selection - 2: Time taken to select the first peg again, measuring sustained attention and readiness.
  Transport Drops - 2: No. of drops during the second transport attempt, evaluating precision and control.
  An increase in moving duration indicates a decline in eye-hand coordination speed.
To determine the effect of EnXtra® and EnXtra® + Caffeine on Sustained attention as assessed by Continuous Performance test (CPT) as compared to placebo and caffeine in acute stage. | Day 0; Day 5; Day 10; Day 15 - 0, 1, 3 & 5 hours ±15 minutes post IP
  This task is primarily designed to measure selective and sustained attention, with some capacity to assess impulsivity to a lesser degree. CPT measures sustained attention and response time. Sustained attention is measured by assessing how well participants can maintain their focus throughout the test. The response time is measured by calculating the average time it takes for a participant to respond to target stimuli. In the CPT, a decline in sustained attention is often reflected in increased response times and greater variability. This can occur as participants become fatigued or distracted over time, leading to slower and less consistent responses.Hence, a long response time may suggest cognitive slowing and/or impairment.
To determine the effect of EnXtra® and EnXtra® + Caffeine on Sustained attention as assessed by Continuous Performance test (CPT) as compared to placebo and caffeine in sub-acute stage. | Day 20 - 0 hours, Day 48 - 1, 3 & 5 hours ±15 minutes post IP
  This task is primarily designed to measure selective and sustained attention, with some capacity to assess impulsivity to a lesser degree. CPT measures sustained attention and response time. Sustained attention is measured by assessing how well participants can maintain their focus throughout the test. The response time is measured by calculating the average time it takes for a participant to respond to target stimuli. In the CPT, a decline in sustained attention is often reflected in increased response times and greater variability. This can occur as participants become fatigued or distracted over time, leading to slower and less consistent responses.Hence, a long response time may suggest cognitive slowing and/or impairment.
To determine the effect of EnXtra® and EnXtra® + Caffeine on Fatigue as assessed by the change in the Samn-Perelli fatigue scale (SPS) compared to placebo and caffeine in acute stage. | Day 0; Day 5; Day 10; Day 15 - 0, 1, 3 & 5 hours ±15 minutes post IP
  SPS is a uni-dimensional 7-point scale that was specifically developed to estimate fatigue in pilots. It is also a 7-point Likert-type scale of subjective fatigue ranging from 1 = "fully alert, wide awake, extremely peppy" to 7 = "completely exhausted, unable to function effectively, ready to drop.
To determine the effect of EnXtra® and EnXtra® + Caffeine on Fatigue as assessed by the change in the Samn-Perelli fatigue scale (SPS) compared to placebo and caffeine in sub-acute stage. | Day 20 - 0 hours, Day 48 - 1, 3 & 5 hours ±15 minutes post IP
  SPS is a uni-dimensional 7-point scale that was specifically developed to estimate fatigue in pilots. It is also a 7-point Likert-type scale of subjective fatigue ranging from 1 = "fully alert, wide awake, extremely peppy" to 7 = "completely exhausted, unable to function effectively, ready to drop.
To determine the safety of EnXtra® and EnXtra® + Caffeine as assessed by the Complete Blood Count - CBC | Screening and Day 48
  The CBC typically includes:
  1. WBC total and differential count (Reference range: 4 - 10 10^3/microlitres)-
  2. erythrogram (RBC count (Reference range: 4.5 - 5.5 10^6/microlitres), determination of hemoglobin (Hb) (Reference range: 12.0 - 17.0 g/dL) and hematocrit (Reference range: 40 - 50 %), and indices calculation (mean corpuscular volume (MCV) (Reference range: 83-101 fL), mean corpuscular hemoglobin (MCH) (Reference range: 27 - 32 pg), mean corpuscular hemoglobin concentration (MCHC) (Reference range: 31.5 - 34.5 g/dL), and red cell distribution width (RDW) (Reference range: 11.6 - 14.0 %) and;
  3. platelet count (Reference range: 7.4 - 11.4 fL) indices calculation
To determine the safety of EnXtra® and EnXtra® + Caffeine as assessed by the Liver Function Tests (LFT) | Screening and Day 48
  The liver function tests (LFT) typically include alanine transaminase (ALT) (Reference range: 9-72 IU/L) and aspartate transaminase (AST) (Reference range: 14-59 IU/L), alkaline phosphatase (ALP) (Reference range: 38-126 U/L). These tests aid in identifying areas of liver damage and, based on the elevation pattern, contribute to forming a differential diagnosis.
To determine the safety of EnXtra® and EnXtra® + Caffeine as assessed by the Kidney Function Tests (KFT) | Screening and Day 48
  The kidney function tests (KFT) typically include serum creatinine (Reference range: 0.5 - 1.4 mg/dL) and blood urea nitrogen (BUN) (Reference range: 7-23 mg/dL). These tests help to evaluate renal function and detect the presence of kidney disease.

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - New Manak Healcare Hospital, Navi Mumbai, Maharashtra
  - Gurukrupa Hospital, Thane, Maharashtra
  - Kalpana Hospital, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: No